CLINICAL TRIAL: NCT02666807
Title: Effects of Oral Ginger Supplementation on NF-KB (Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells) in Peripheral Blood Mononuclear Cells (PBMC) and Glycemic and Lipid Profiles in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Ginger Supplementation on NF-KB in Peripheral Blood Mononuclear Cells in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Niaz Mohammadzadeh Honarvar, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: TehranUMS
Record Dates: First submitted 2016-01-10; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: NF-κB; Ginger
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ginger extract; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger (Experimental): Ginger (Zingiber officinale Roscoe) 500 mg capsules (2000 mg per day) by mouth twice daily (BID) for 10 weeks
  Interventions: Dietary Supplement: Ginger
- Placebo (Placebo Comparator): Placebo matching with ginger 0 mg capsules by mouth twice daily (BID) for 10 weeks Placebo twice daily
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Ginger — Ginger 500 mg capsules (2000 mg per day) by mouth twice daily (BID) for 10 weeks
  Other Names: Zingiber officinale Roscoe
  Arms: Ginger
Dietary Supplement: placebo — Placebo matching with ginger 0 mg capsules by mouth twice daily (BID) for 10 weeks
  Other Names: wheat flour capsules
  Arms: Placebo

SUMMARY:
This study evaluates the effect of ginger on NF-KB level in Peripheral Blood Mononuclear Cells in type 2 diabetic patients. Half of patients will receive ginger, while the other half will receive placebo.

DETAILED DESCRIPTION:
ginger is a plant with lots of phytochemicals which have antioxidant effects. It reduces the NF-KB levels in the cells because of its antioxidant effects. It can reduces insulin resistance as a result of NF-KB reduction in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 of diabetes diagnosed for 1 to 10 years
* age 30-60 years
* BMI = 18.5-35 kg/m*m
* treatment with Metformin or Glibenclamide

Exclusion Criteria:

* Treatment with insulin
* Weight loss more than 10% in 6 months
* Treatment with TZDs (thiazolidinediones)
* Pregnancy and breast feeding
* Smoking and alcohol consumption
* Multivitamin-mineral and polyphenols and omega-3 and 6 supplementation in the last 3 months and during study
* Ginger supplementation and herbal medicines
* Anticoagulation consumption such as heparin and warfarin
* NSAIDs such as diclofenac and salicylate drugs such as aspirin, corticosteroids such as prednisone consumption during 1 month ago and during the study
* Infectious and inflammatory diseases such as rheumatoid arthritis
* Impaired hepatic, renal and gastrointestinal function
* Cancer
* Currently suffering from acute illness that needs medical treatment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in NF-KB at 10 weeks | Baseline and 10 weeks

SECONDARY OUTCOMES:
Change from Baseline in FBS (mg/dl) at 10 weeks | Baseline and 10 weeks
  FBS (Fasting Blood sugar) (mg/dl)
Change from Baseline in HDL-C (mg/dl) at 10 weeks | Baseline and 10 weeks
  HDL-C (High Density Lipoprotein) (mg/dl)
Change from Baseline in LDL-C (mg/dl) at 10 weeks | Baseline and 10 weeks
  LDL-C (Low Density Lipoprotein) (mg/dl)
Change from Baseline in Total-C (mg/dl) at 10 weeks | Baseline and 10 weeks
  Total-C (Total Cholesterol) (mg/dl)
Change from Baseline in TG (mg/dl) at 10 weeks | Baseline and 10 weeks
  TG (Triacylglycerol) (mg/dl)
Change from Baseline in Hb A1C at 10 weeks | Baseline and 10 weeks
  Hb A1C (Glycated hemoglobin)
Change from Baseline in insulin (µlU/ml) at 10 weeks | Baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Saedisomeolia, Prof.assoc, Study Director — Tehran University of Medical Sciences; Motahare Makhdoomiarzati, Msc student, Principal Investigator — Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jung HW, Yoon CH, Park KM, Han HS, Park YK. Hexane fraction of Zingiberis Rhizoma Crudus extract inhibits the production of nitric oxide and proinflammatory cytokines in LPS-stimulated BV2 microglial cells via the NF-kappaB pathway. Food Chem Toxicol. 2009 Jun;47(6):1190-7. doi: 10.1016/j.fct.2009.02.012. Epub 2009 Feb 20. PMID 19233241
- [Result] Ali BH, Blunden G, Tanira MO, Nemmar A. Some phytochemical, pharmacological and toxicological properties of ginger (Zingiber officinale Roscoe): a review of recent research. Food Chem Toxicol. 2008 Feb;46(2):409-20. doi: 10.1016/j.fct.2007.09.085. Epub 2007 Sep 18. PMID 17950516
- [Result] Li XH, McGrath KC, Tran VH, Li YM, Duke CC, Roufogalis BD, Heather AK. Attenuation of Proinflammatory Responses by S-[6]-Gingerol via Inhibition of ROS/NF-Kappa B/COX2 Activation in HuH7 Cells. Evid Based Complement Alternat Med. 2013;2013:146142. doi: 10.1155/2013/146142. Epub 2013 Jun 16. PMID 23843863
- [Result] Ogawa Y, Yamaguchi K, Tanaka T, Morozumi M, Kitagawa R. [Evaluation of the enzymatic method using oxalate oxidase for urinary oxalate assay]. Hinyokika Kiyo. 1987 Dec;33(12):1951-4. Japanese. PMID 3448918